CLINICAL TRIAL: NCT03006640
Title: Subcutaneous NTG for US Radial Artery Cannulation
Acronym: NTG-US-art
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AlRefaey Kandeel (Other)
Responsible Party: Sponsor-Investigator, AlRefaey Kandeel, Dr, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Refa-NTG-art
Record Dates: First submitted 2016-12-27; First posted 2016-12-30 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Placebo Comparator)
  Interventions: Drug: Subcutaneous saline
- NTG group (Active Comparator)
  Interventions: Drug: Subcutaneous nitroglycrin

INTERVENTIONS:
Drug: Subcutaneous nitroglycrin — In both groups, a 1 ml filled insulin syringe is delivered to a blinded operator who infiltrated it subcutaneously over 1 cm along the radial artery course. In the NTG group, the syringe contains 200 µg of NTG while in control group the syringe is filled with saline
  Arms: NTG group
Drug: Subcutaneous saline — In both groups, a 1 ml filled insulin syringe is delivered to a blinded operator who infiltrated it subcutaneously over 1 cm along the radial artery course. In the NTG group, the syringe contains 200 µg of NTG while in control group the syringe is filled with saline
  Arms: Control group

SUMMARY:
Clinicians are increasingly dealing with morbid obese patients. In morbid obese patients, difficult sampling and problems encountered with noninvasive blood pressure monitoring makes arterial cannulation an essential skill in many situations like surgeries or trans-radial procedures for coronary or carotid interventions.

Radial artery has been preferred over other sites for arterial cannulation due to low incidence of bleeding, better hemostats, more comfort, and immediate ambulation. sm In this study, subcutaneous nitroglycerin will be used to facilitate radial artery cannulation aiming to decrease insertion time, increase success rate and decrease related complications

ELIGIBILITY:
Inclusion Criteria:

* morbid obese indicated for radial artery cannuulation

Exclusion Criteria:

* +ve allen test peripheral arterial disease refusal

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Success rate | 24 hours after surgery

IPD SHARING:
Plan to Share IPD: Undecided